CLINICAL TRIAL: NCT05061316
Title: The Gut Microbiome As an Indicator of Readiness for Head & Neck Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Carissa M Thomas, MD PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007821
Record Dates: First submitted 2021-08-30; First posted 2021-09-29 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer of Head and Neck; Nutrition Aspect of Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition intervention group (Experimental): Participants will receive Nestlé Impact Advanced Recovery Immunonutrition two times daily for 5 days leading up to the date of surgery. Nestlé Impact Advanced Recovery will be administered either orally or through a feeding tube.
  Interventions: Dietary Supplement: Nestlé Impact Advanced Recovery

INTERVENTIONS:
Dietary Supplement: Nestlé Impact Advanced Recovery — Immunonutrition drink that helps support the immune system: reduces risk of prolonged hospital stay and complications after surgery.

SUMMARY:
The purpose of this study is to understand how a pre-operative nutritional intervention alters the gut microbiome and improves outcomes after major head and neck cancer surgery.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) arises from the mucosal lining of the upper aerodigestive system. Tumor-associated pain and physical obstruction from the tumor can impair a patient's ability to eat, and this combined with the catabolic nature of cancer leads to significant weight loss.HNC patients have a high burden of moderate to severe malnutrition and cachexia with a rate of approximately 40%, and malnourishment at the time of HNC diagnosis is associated with poor survival. In addition, these malnourished patients have longer post-operative hospital length of stay, increased post-operative complications including infection, delayed wound healing, muscle weakness, impaired cardiac and respiratory symptoms, reduced response to adjuvant treatment, and decreased quality of life. Inflammation increases the risk of malnutrition and may play a role in the suboptimal response to certain nutrition interventions.

Changes in diversity and relative abundance of gut bacteria in malnourished patients with head and neck cancer after a pre-operative nutrition intervention will be determined. Post-operative outcomes including wound complications, other surgical and medical complications, hospital length of stay, unintended readmission within 30 days and mortality after a pre-operative nutrition intervention will be recorded and compared to a historic control. Finally, changes in known markers of nutritional status (albumin, prealbumin, c-reactive protein (CRP), transferrin, thyroid stimulating hormone (TSH), comprehensive metabolic panel (CMP), and complete blood count (CBC)) and systemic inflammatory markers (Interleukin (IL)-1β, IL-6, IFNγ, TNF, IL-2, IL-4, IL-10, IL-12, IL-17) will be measured after a pre-operative nutrition intervention. The pre-operative nutrition intervention is Nestlé Impact Advanced Recovery Immunonutrition administered orally or through a feeding tube two times daily for 5 days leading up to the date of surgery (day -5 to -1). Nestlé Impact Advanced Recovery provides 280kcal, 11g total fat, 20g carbohydrates, and 26g protein per unit (250mL). In addition, it is enriched with L-arginine and omega-3 fatty acids, two components found to be essential for the beneficial effect of immunonutrition in a systematic review.

Immunonutrition is a specially formulated diet that contains nutrients to modulate inflammation. Pre-operative nutrition interventions with immunonutrition have demonstrated a decrease in post-operative complications (35% vs 50%, p=0.034) and unplanned readmissions and shortened hospital stays (17 vs 6 days, p<0.001) in patients with HNC. Studies have shown that dietary interventions can improve wound healing and post-operative survival. Currently, nothing is known about the composition of the gut microbiome in malnourished patients with HNC and how that composition changes with an immunonutrition intervention. There is evidence that remote tissue healing is influenced by the gut microbiome. In mice undergoing a pre-operative nutrition intervention, there is a shift in the gut microbiome composition from Proteobacteria and Firmicutes to Bacteroidetes, which produce metabolites that impact the systemic immune system.

The study hypothesis is the gut microbiome can serve as a marker of readiness for major surgery after a pre-operative nutrition intervention in patients with HNC. The investigators aim to treat malnourished patients with HNC with immunonutrition and examine changes in the gut microbiome composition to define a gut microbiome associated with decreased post-operative complications, improved markers of nutritional status, and decreased markers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18+)
* Male or female
* Diagnosis of head and neck cancer that will be treated with major surgery
* Major surgeries included will be any free flap reconstruction, any regional flap reconstruction (including pec major, submental flap, and supraclavicular artery island flap), oral composite resection, oropharyngectomy, total laryngectomy, cutaneous malignancy if it includes a free flap or regional flap reconstruction, parotidectomy if it includes a free flap or regional flap reconstruction, maxillectomy with or without orbital exenteration, lateral temporal bone resection, and/or a radical neck dissection if it includes a free flap or regional flap reconstruction
* Diagnosis of moderate (Stage B) or severe (Stage C) malnutrition, based on the patient-generated subjective global assessment (PG-SGA)
* Ability to speak and comprehend English
* Ability to consent for themselves

Exclusion Criteria:

* Age less than 18 years
* Inability to speak and comprehend English
* Inability to consent for themselves
* Pregnancy
* Allergy to fish oil or fish
* Gastrointestinal disorders (IBD, colon or rectal cancer, previous colon or small intestine resection)
* Autoimmune disorders requiring medication
* Chronic immunosuppression (i.e., transplant patients)
* Leukemia
* Stage III or higher Chronic Kidney Disease (CKD)
* Cirrhosis
* Pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Define changes in the gut microbiome in malnourished patients with head and neck cancer after a pre-operative nutrition intervention via analyses of stool samples. | Baseline - 6 months
  Stool samples will be collected prior to the nutrition intervention and after completing 5 days of intervention. Stool samples will be processed and sequenced for 16S microbiome analysis. The composition of the gut microbiome will be compared before and after the immunonutrition intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carissa M. Thomas, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No